CLINICAL TRIAL: NCT01714687
Title: Comparison of Balloon Sinuplasty In-Office Versus Medical Management for Recurrent Acute Sinusitis Patients: A Randomized Controlled Study (CABERNET)
Brief Title: Comparison of Balloon Sinuplasty In-Office Versus Medical Management for Recurrent Acute Sinusitis Patients (CABERNET)
Acronym: CABERNET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPR005030
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Recurrent Acute Rhinosinusitis
MeSH Terms: interventions — Nutrition Therapy; Practice Management, Medical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- balloon sinus dilation (Active Comparator): Balloon sinus dilation will be conducted in-office under local anesthesia.
  Interventions: Device: balloon sinus dilation; Other: medical therapy
- medical therapy (Active Comparator): Medical therapy as needed per subject's specific disease and as determined by the investigators' clinical judgment.
  Interventions: Other: medical therapy

INTERVENTIONS:
Device: balloon sinus dilation
  Other Names: balloon sinuplasty
  Arms: balloon sinus dilation
Other: medical therapy
  Other Names: medical management

SUMMARY:
This post-market study aims to compare health outcomes for Recurrent Acute Rhinosinusitis (RARS) patients treated with balloon sinus dilation (BSD) versus medical management alone.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or greater
* diagnosis of recurrent acute rhinosinusitis
* suitable candidate for office-based procedure
* willing and able to read and sign informed consent and remain compliant with protocol and study procedures
* able to read and understand English

Exclusion Criteria:

* diagnosis of chronic rhinosinusitis
* prior sinus surgery
* physician determined need for ancillary procedures
* known immune deficiency, ciliary dysfunction and/or autoimmune disease
* clinically significant illness that may interfere with evaluation of the study
* participation in clinical studies 6 months prior to study participation
* pregnant or lactating females

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2016-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Sikand, MD, Principal Investigator — Ear Nose and Throat Consultants of Nevada; Ford Albritton, MD, Principal Investigator — Texas Institute for Sinus & Respiratory Disease
Locations (5):
- United States (5):
  - Birmingham, Alabama
  - Atlanta, Georgia
  - Las Vegas, Nevada
  - Dallas, Texas
  - McKinney, Texas

IPD SHARING:
Plan to Share IPD: Yes
Publication planned in the future

RESULTS

PARTICIPANT FLOW:
Groups:
- Balloon Sinus Dilation: Subjects treated with balloon sinus dilation
- Medical Therapy: Subjects treated with medical therapy as needed per the subject's specific disease and as determined by the investigator's clinical judgement.
Period: Overall Study
Arm/Group | Balloon Sinus Dilation | Medical Therapy
Started | 29 | 30
Completed | 26 | 26
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Balloon Sinus Dilation | Medical Therapy | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (10.0) | 43.8 (9.7) | 45.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 23 | 28 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: CSS Total Score Change From Baseline to 24 Week Visit
Description: The Chronic Sinusitis Survey (CSS) is a 6 question, duration-based survey to evaluate surgical outcomes for CRS patients. The CSS asks three questions about symptoms and three questions about medication usage and yields a symptom subscore, a medication subscore, and a total score. Scale values include "0 Weeks" (minimum), "1-2 Weeks", "3-4 Weeks", "5-6 Weeks", and "7-8 Weeks" (maximum).
  The severity of symptoms is scored 0 (none) to 4 (severe), and a total score is calculated from 0 (worst) to 100 (best). Subscores are averaged to calculate a total score. Higher score indicates better outcomes.
  The Primary Endpoint is the comparison of change in total CSS score over 24 weeks for subjects randomized to BSD versus medical management only.
  Change is assessed by using the Mean Change for the CSS total score at 24 weeks compared to baseline. (24-week CSS total score minus Baseline CSS total score).
  Higher score indicates greater improvement.
Time Frame: 24 Week Visit
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Balloon Sinus Dilation | Medical Therapy
Number analyzed (Participants) | 29 | 30
scores on a scale | 37.3 (24.4) | 21.8 (29.0)

2. Secondary Outcome: CSS Sub-score Changes From Baseline Over 48 Weeks, and CSS Total Score Over 48 Weeks
Description: The Chronic Sinusitis Survey (CSS) is a 6 question, duration-based survey ("0 Weeks" (minimum) to "7-8 Weeks" (maximum)) used to evaluate surgical outcomes for CRS patients. The CSS asks 3 questions each about symptoms and medication usage, yielding a symptom subscore, a medication subscore, and a total score. The symptom-based section contains pain or pressure, nasal congestion or difficulty to breathe through the nose, and rhinorrhea or postnasal drip. The medication-based section contains: antibiotics, prescription nasal sprays, and sinus medications in pill form. The severity of symptoms is scored 0 (none) to 4 (severe), and a total score is calculated from 0 (worst) to 100 (best). The Secondary Endpoint is the comparison of change as measured by average CSS medication and sinusitis symptom sub-scores over 24 and 48 weeks, and average total CSS score over 48 weeks for subjects randomized to BSD versus medical management. Higher score indicates greater improvement.
Time Frame: 8, 16, 24, 32, 40, and 48 Weeks
Population: All available date for each follow-up visit is presented.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Balloon Sinus Dilation | Medical Therapy
Number analyzed (Participants) | 29 | 30
scores on a scale
  CSS Symptom Sub-score Change at Procedure: number analyzed (Participants) | 28 | 30
  CSS Symptom Sub-score Change at Procedure | 3.9 (19.4) | -7.5 (21.4)
  CSS Symptom Sub-score Change at Week 8: number analyzed (Participants) | 28 | 28
  CSS Symptom Sub-score Change at Week 8 | 39.6 (33.7) | 24.1 (39.6)
  CSS Symptom Sub-score Change at Week 16: number analyzed (Participants) | 27 | 28
  CSS Symptom Sub-score Change at Week 16 | 46.3 (32.0) | 30.1 (38.9)
  CSS Symptom Sub-score Change at Week 24: number analyzed (Participants) | 26 | 27
  CSS Symptom Sub-score Change at Week 24 | 48.7 (28.7) | 27.2 (40.1)
  CSS Symptom Sub-score Change at Week 32: number analyzed (Participants) | 24 | 8
  CSS Symptom Sub-score Change at Week 32 | 45.8 (33.8) | 35.4 (24.7)
  CSS Symptom Sub-score Change at Week 40: number analyzed (Participants) | 23 | 7
  CSS Symptom Sub-score Change at Week 40 | 52.9 (32.7) | 29.8 (22.0)
  CSS Symptom Sub-score Change at Week 48: number analyzed (Participants) | 22 | 6
  CSS Symptom Sub-score Change at Week 48 | 53.8 (24.6) | 33.3 (25.9)
  CSS Medication Sub-score Change at Procedure: number analyzed (Participants) | 28 | 30
  CSS Medication Sub-score Change at Procedure | -1.5 (17.1) | -7.0 (17.4)
  CSS Medication Sub-score Change at Week 8: number analyzed (Participants) | 28 | 28
  CSS Medication Sub-score Change at Week 8 | 27.7 (27.4) | 12.2 (22.9)
  CSS Medication Sub-score Change at Week 16: number analyzed (Participants) | 27 | 28
  CSS Medication Sub-score Change at Week 16 | 25.0 (27.6) | 12.2 (22.5)
  CSS Medication Sub-score Change at Week 24: number analyzed (Participants) | 26 | 27
  CSS Medication Sub-score Change at Week 24 | 26.0 (26.6) | 16.4 (24.0)
  CSS Medication Sub-score Change at Week 32: number analyzed (Participants) | 24 | 8
  CSS Medication Sub-score Change at Week 32 | 35.1 (23.2) | 26.0 (32.0)
  CSS Medication Sub-score Change at Week 40: number analyzed (Participants) | 23 | 7
  CSS Medication Sub-score Change at Week 40 | 37.0 (24.5) | 30.9 (31.1)
  CSS Medication Sub-score Change at Week 48: number analyzed (Participants) | 22 | 6
  CSS Medication Sub-score Change at Week 48 | 30.7 (22.0) | 27.8 (30.6)
  Total CSS Change Change at Procedure: number analyzed (Participants) | 28 | 30
  Total CSS Change Change at Procedure | 1.2 (14.3) | -7.2 (16.1)
  Total CSS Change Change at Week 8: number analyzed (Participants) | 28 | 28
  Total CSS Change Change at Week 8 | 33.6 (27.5) | 18.2 (26.4)
  Total CSS Change Change at Week 16: number analyzed (Participants) | 27 | 28
  Total CSS Change Change at Week 16 | 35.6 (24.9) | 21.1 (27.1)
  Total CSS Change Change at Week 24: number analyzed (Participants) | 26 | 27
  Total CSS Change Change at Week 24 | 37.3 (24.4) | 21.8 (29.0)
  Total CSS Change Change at Week 32: number analyzed (Participants) | 24 | 8
  Total CSS Change Change at Week 32 | 40.5 (22.9) | 30.7 (24.3)
  Total CSS Change Change at Week 40: number analyzed (Participants) | 23 | 7
  Total CSS Change Change at Week 40 | 44.9 (22.5) | 30.4 (24.0)
  Total CSS Change Change at Week 48: number analyzed (Participants) | 22 | 6
  Total CSS Change Change at Week 48 | 42.2 (17.9) | 30.6 (24.2)

3. Secondary Outcome: RSDI Total and Sub-score Changes From Baseline Over 48 Weeks
Description: The Rhinosinusitis Disability Index (RSDI) is a 30-question survey which includes 3 individual subscales to measure physical, functional, and emotional scores as well as a total score. There is no specified recall period. Scale values include "Never" (minimum), "Almost Never", "Sometimes", "Almost Always", "Always" (maximum).
  RSDI scores range from 0 to 120. Subscores are averaged to calculate a total score. Higher score indicates increased impact of sinus disease.
  The Secondary Endpoint is comparison of change in patient-reported QOL as measured by RSDI total, physical, functional, and emotional sub-scores at 8, 24 and 48 weeks for subjects randomized to BSD versus medical management.
  Lower score indicates greater improvement (decreased impact of sinus disease).
Time Frame: 8, 24, and 48 Weeks
Population: All available data for each follow-up visit is presented.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Balloon Sinus Dilation | Medical Therapy
Number analyzed (Participants) | 29 | 30
scores on a scale
  RSDI Total Change at Procedure: number analyzed (Participants) | 28 | 30
  RSDI Total Change at Procedure | -1.0 (13.4) | 2.5 (9.0)
  RSDI Total Change at Week 8: number analyzed (Participants) | 28 | 28
  RSDI Total Change at Week 8 | -32.9 (26.8) | -17.9 (30.9)
  RSDI Total Change at Week 24: number analyzed (Participants) | 26 | 27
  RSDI Total Change at Week 24 | -35.6 (28.2) | -18.7 (27.4)
  RSDI Total Change at Week 48: number analyzed (Participants) | 22 | 6
  RSDI Total Change at Week 48 | -36.9 (21.1) | -17.2 (14.9)
  RSDI Physical Sub-score Change at Procedure: number analyzed (Participants) | 28 | 30
  RSDI Physical Sub-score Change at Procedure | -1.8 (5.7) | 0.5 (3.4)
  RSDI Physical Sub-score Change at Week 8: number analyzed (Participants) | 28 | 28
  RSDI Physical Sub-score Change at Week 8 | -14.5 (11.2) | -8.6 (12.4)
  RSDI Physical Sub-score Change at Week 24: number analyzed (Participants) | 26 | 27
  RSDI Physical Sub-score Change at Week 24 | -15.4 (10.8) | -9.1 (12.1)
  RSDI Physical Sub-score Change at Week 48: number analyzed (Participants) | 22 | 6
  RSDI Physical Sub-score Change at Week 48 | -15.1 (9.3) | -8.5 (6.3)
  RSDI Emotional Sub-score Change at Procedure: number analyzed (Participants) | 28 | 30
  RSDI Emotional Sub-score Change at Procedure | 1.2 (5.0) | 1.8 (3.8)
  RSDI Emotional Sub-score Change at Week 8: number analyzed (Participants) | 28 | 28
  RSDI Emotional Sub-score Change at Week 8 | -8.6 (8.9) | -4.0 (11.2)
  RSDI Emotional Sub-score Change at Week 24: number analyzed (Participants) | 26 | 27
  RSDI Emotional Sub-score Change at Week 24 | -9.8 (9.2) | -3.9 (9.1)
  RSDI Emotional Sub-score Change at Week 48: number analyzed (Participants) | 22 | 6
  RSDI Emotional Sub-score Change at Week 48 | -10.4 (7.3) | -3.7 (5.6)
  RSDI Functional Sub-score Change at Procedure: number analyzed (Participants) | 28 | 30
  RSDI Functional Sub-score Change at Procedure | -0.4 (5.2) | 0.2 (3.9)
  RSDI Functional Sub-score Change at Week 8: number analyzed (Participants) | 28 | 28
  RSDI Functional Sub-score Change at Week 8 | -9.8 (8.2) | -5.3 (9.4)
  RSDI Functional Sub-score Change at Week 24: number analyzed (Participants) | 26 | 27
  RSDI Functional Sub-score Change at Week 24 | -10.4 (9.6) | -5.7 (7.9)
  RSDI Functional Sub-score Change at Week 48: number analyzed (Participants) | 22 | 6
  RSDI Functional Sub-score Change at Week 48 | -11.4 (7.1) | -5.0 (4.9)

4. Secondary Outcome: Medication Usage at 24 and 48 Weeks
Description: Comparison of medication usage at 24 and 48 weeks (days oral antibiotics, oral steroids, topical intranasal steroid sprays, and 'atypical' topical steroids (drops or respules)) for subjects randomized to BSD versus medical management.
Time Frame: 24 Weeks and 48 Weeks
Population: All available data for each follow-up visit is presented.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Balloon Sinus Dilation | Medical Therapy
Number analyzed (Participants) | 29 | 30
Days
  Oral Antibiotics at 24 Week Visit: number analyzed (Participants) | 26 | 27
  Oral Antibiotics at 24 Week Visit | 0.7 (2.3) | 2.9 (6.6)
  Oral Antibiotics at 48 Week Visit: number analyzed (Participants) | 22 | 5
  Oral Antibiotics at 48 Week Visit | 0.5 (2.1) | 2.0 (3.1)
  Injected Antibiotics at 24 Week Visit: number analyzed (Participants) | 26 | 27
  Injected Antibiotics at 24 Week Visit | 0.0 (0.0) | 0.0 (0.0)
  Injected Antibiotics at 48 Week Visit: number analyzed (Participants) | 22 | 5
  Injected Antibiotics at 48 Week Visit | 0.0 (0.2) | 0.0 (0.0)
  Oral Steroids at 24 Week Visit: number analyzed (Participants) | 26 | 27
  Oral Steroids at 24 Week Visit | 0.6 (2.8) | 1.0 (3.1)
  Oral Steroids at 48 Week Visit: number analyzed (Participants) | 22 | 5
  Oral Steroids at 48 Week Visit | 0.7 (2.4) | 0.0 (0.0)
  Nasal Steroid Sprays at 24 Week Visit: number analyzed (Participants) | 26 | 27
  Nasal Steroid Sprays at 24 Week Visit | 10.5 (19.0) | 21.5 (24.0)
  Nasal Steroid Sprays at 48 Week Visit: number analyzed (Participants) | 21 | 5
  Nasal Steroid Sprays at 48 Week Visit | 10.3 (19.8) | 24.0 (29.4)

5. Secondary Outcome: Unscheduled Medical Care Visits Due to Sinusitis
Description: Comparison of unscheduled medical care visits due to sinusitis at 24 and 48 weeks for subjects randomized to BSD versus medical management.
Time Frame: 24 Weeks and 48 Weeks
Population: All available data for each follow-up visit is presented.
Measure: Mean (Standard Deviation); unit: Medical care visits
Arm/Group | Balloon Sinus Dilation | Medical Therapy
Number analyzed (Participants) | 29 | 30
Medical care visits
  Sinus-related visits through 24 weeks: number analyzed (Participants) | 26 | 27
  Sinus-related visits through 24 weeks | 0.2 (0.8) | 0.9 (1.3)
  Sinus-related visits through 48 Weeks: number analyzed (Participants) | 22 | 5
  Sinus-related visits through 48 Weeks | 0.2 (0.9) | 0.2 (0.4)

6. Secondary Outcome: Sinus Infections and Sinus Severity - Part 1
Description: Comparison of number of post-enrollment sinus infections for subjects randomized to BSD versus medical management.
Time Frame: 24 Weeks and 48 Weeks
Population: All available data for each follow-up visit is presented.
Measure: Mean (Standard Deviation); unit: Sinus Infections
Arm/Group | Medical Therapy | Balloon Sinus Dilation
Number analyzed (Participants) | 30 | 29
Sinus Infections
  Sinus infections thru 24 wks: number analyzed (Participants) | 26 | 27
  Sinus infections thru 24 wks | 0.2 (0.4) | 0.9 (0.9)
  Sinus infections thru 48 wks: number analyzed (Participants) | 22 | 5
  Sinus infections thru 48 wks | 0.2 (0.4) | 0.4 (0.5)

7. Secondary Outcome: Sinus Infections and Sinus Severity - Part 2
Description: Comparison of patient-reported sinus infection severity for subjects randomized to BSD versus medical management.
Time Frame: 24 Weeks
Population: All available data for each follow-up visit is presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Therapy | Balloon Sinus Dilation
Number analyzed (Participants) | 30 | 29
Participants
  Severity of Sinus Symptoms thru 24 wks: number analyzed (Participants) | 26 | 27
  Severity of Sinus Symptoms thru 24 wks: Improved or No Sinus Infection | 25 | 16
  Severity of Sinus Symptoms thru 24 wks: No Change | 1 | 10
  Severity of Sinus Symptoms thru 24 wks: Worse | 0 | 1
  Severity of Sinus Infections thru 24 wks: number analyzed (Participants) | 26 | 27
  Severity of Sinus Infections thru 24 wks: Improved or No Sinus Infection | 25 | 18
  Severity of Sinus Infections thru 24 wks: No Change | 1 | 8
  Severity of Sinus Infections thru 24 wks: Worse | 0 | 1

8. Secondary Outcome: Frequency of Second Procedure
Description: Frequency of second procedure, ie the number of medical management subjects (sham arm) electing cross-over procedure.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Therapy
Number analyzed (Participants) | 30
Participants | 18

9. Secondary Outcome: Return to Normal Activity
Description: Days until return to normal activity (RTNA) assessed at 2 weeks post-procedure
Time Frame: 2 week
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Balloon Sinus Dilation | Medical Therapy
Number analyzed (Participants) | 29 | 30
Days | 1.8 (1.6) | 1.3 (1.3)

ADVERSE EVENTS:
Arm/Group | Balloon Sinus Dilation | Medical Therapy
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/30
Other Adverse Events (participants affected / at risk) | 17/29 | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Sinus Dilation (N=29) | Medical Therapy (N=30)
Facial Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Sinus Dilation (N=29) | Medical Therapy (N=30)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 2 (3) | 10 (18)
Upper Respiratory Infection (Infections and infestations) | 3 (3) | 7 (7)
Dental abcess (Infections and infestations) | 0 (0) | 1 (1)
Hyposmia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia, aspiration (Infections and infestations) | 1 (1) | 0 (0)
Cervical Lymphadenopathy (Immune system disorders) | 1 (1) | 0 (0)
Eustachian Tube Dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Infertility (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hernia, abdominal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mononucleosis (Infections and infestations) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nodules of Vocal Code (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Migraine, ocular (Nervous system disorders) | 1 (1) | 0 (0)
Poison Ivy rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthritis, Psoriatic (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhinitis Medicamentosa (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (3) | 1 (1)
Vasovagal Reaction (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days